CLINICAL TRIAL: NCT03463239
Title: Phase 1 Pilot Study of Bioengineered Penile Tissue Constructs in Subjects With Irreversibly Damaged Penile Corpora
Brief Title: Bioengineered Penile Tissue Constructs for Irreversibly Damaged Penile Corpora
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00046975
Record Dates: First submitted 2018-02-18; First posted 2018-03-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-03

CONDITIONS: Urologic Diseases; Male Urogenital Diseases; Penile Diseases; Corpus Callosum Malformation; Corpora Cavernosa; Inflammation; Trauma Injury
Keywords: Autologous tissue engineered corpora
MeSH Terms: conditions — Urologic Diseases; Male Urogenital Diseases; Penile Diseases; Agenesis of Corpus Callosum; Inflammation; Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous tissue engineered corpora (Experimental): All subjects enrolled will undergo a corpora cavernosum biopsy. Endothelial and smooth muscle cells will be isolated and expanded, then seeded onto a scaffold that will later be implanted into the subject.
  Interventions: Biological: Autologous tissue engineered corpora

INTERVENTIONS:
Biological: Autologous tissue engineered corpora — penile tissue construct

SUMMARY:
The primary objective of this clinical trial is to evaluate the safety of autologous engineered corpora cavernosa + albuginea constructs for treatment of complex penile deformities. Autologous endothelial and smooth muscle cells obtained from enrolled subjects' corpora cavernosa biopsy sample, will be culture expanded in vitro and used to seed decellularized corpora cavernosa + albuginea obtained from cadaveric-donors to create autologous bioengineered corpora cavernosa/albuginea constructs for repair of damaged penile tissues.

DETAILED DESCRIPTION:
Damage to penile tissue due to infection, inflammation or trauma often leads to structural deformity that may result in loss of sexual function that can profoundly affect quality of life. Traumatic injuries in civilians and battlefield related injuries in soldiers often require reconstructive procedures to restore the anatomy and functionality of the penis. However, these procedures are often limited by poor availability of functionally intact penile tissue. Various penile reconstructive procedures, such as penile prostheses and autograft implantation have been attempted. While cosmetic appearance may be improved, restoration of spontaneous and natural erectile function is usually not achieved. This is often due to critical defect of the corpora cavernosa, which are responsible for erectile function. Recently, the concept of a tissue engineering-based therapy has been proposed for reconstructing damaged penile corporal tissue.

The primary objective of this Armed Forces Institute for Regeneration Medicine (AFIRM II) sponsored clinical trial is to evaluate the safety of autologous engineered corpora cavernosa + albuginea constructs for treatment of complex penile deformities. The proposed study design is a prospective non-randomized and uncontrolled, multi-center investigation. Autologous endothelial and smooth muscle cells obtained from enrolled participants' corpora cavernosa biopsy sample, will be culture expanded in vitro and used to seed decellularized corpora cavernosa + albuginea obtained from cadaveric-donors to create autologous bioengineered corpora cavernosa/albuginea constructs for repair of damaged penile tissues.

A total of ten male patients, referred for the treatment of damages of albuginea and/or corpora cavernosum without concurrent urethral injury will be recruited for this study. The estimated duration of the study for each subject following treatment is 36 months. The study team anticipates a duration of approximately 48 to 60 months to complete all enrollment and follow up. Enrolled participants will undergo a corporal tissue biopsy as an out-patient surgical procedure. Autologous corporal smooth muscle cells and corporal endothelial cells will be isolated and then seeded on cadaveric decellularized corporal bodies. Approximately 3-4 weeks later, the engineered construct including corporal tissue with attached tunica will be transplanted into the surgically prepared site of penile injury. Participants will be followed through 36 months post-implantation to monitor for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18-60 years.
2. Acquired structural abnormalities of the corpora cavernosum secondary to trauma, infection, inflammation, or fibromatosis. These abnormalities will be diagnosed by clinical examination, and/or ultrasound, and/or computerized tomography.
3. Stable abnormalities - at least 6 months with no pain or changes in deformity.
4. At least one failed attempt at management by conventional approaches at least 6 months prior to enrollment
5. Deformities less than 5 cm in length.
6. Written informed consent obtained prior to participation in the study.
7. Patients must be available for all follow up visits.
8. Ability to speak English.

Exclusion Criteria:

1. Presence of untreated or incompletely treated urinary tract infection at the time of biopsy.
2. Uncontrolled bleeding disorder or patients with a platelet count less than 50,000, hemophilia or patients routinely receiving blood products for bleeding disorders.
3. Serum creatinine > 2.0 mg/dl or evidence of progressive renal disease.
4. ALT or AST value >1.5 times the upper limit of normal.
5. Albumin < 3.0 g/dL.
6. Serum direct bilirubin >0.3 mg/dL OR total bilirubin > 1.4 mg/dL
7. BM I>40 kg/m2
8. Uncontrolled diabetes with HbA1C>9%. (Subjects with controlled diabetes must be under care of diabetologist with treatment goals consistent with ADA criteria).
9. Unstable cardiac disorders within the past 6 months including angina, abnormal ECG, history of cardiac arrest, surgery and/or other interventional procedure.
10. Unstable pulmonary disorders within the past 6 months including dyspnea on exertion, chronic productive cough, pneumonia, hemoptysis, asthma requiring nebulized therapy.
11. Active tuberculosis (TB) requiring treatment in the past 3 years. Subjects with a current positive (≥5 mm induration for high-risk subjects; otherwise ≥10 mm of induration) purified protein derivative (PPD) test are excluded unless they have completed a full course of treatment for latent TB and have a negative chest x-ray film at enrollment.
12. Known to be colonization with either methicillin-resistant Staphylococcus aureus (MRSA) or vancomycin-resistant Enterococcus (VRE), or gentamicin-resistant organisms.
13. Immunocompromised subjects or subjects receiving immunosuppressive agents.
14. Any history of alcohol and/or drug abuse.
15. Documented history of, or positive result of HIV, Hepatitis B or C, or any infectious disease. External signs, sequelae, or positive serology of sexually transmitted disease (including HPV). Patients with a history of systemic conditions, including but not limited to HIV, diabetes and chronic liver disease (including Hepatitis B or C), that the Investigator believes may jeopardize the safety of the patient to participate in the study.
16. Concurrent participation in any other clinical investigation during the period of this investigation. Patients who have been treated with any other investigational drug or participated in any investigational study within 30 days prior to enrollment in this study.
17. Any circumstance in which the investigator deems participation in the study is not in the subject's best interest.
18. Inability to participate in all necessary study activities due to physical or mental limitations.
19. Inability or unwillingness to return for all required follow-up visits, for instance life expectancy < 1 year, or subject who knows they will be moving out of the country and unable to return for follow-up visits.
20. Inability or unwillingness to sign informed consent.
21. Patients requiring concomitant use of or treatment with immunosuppressive agents
22. Patients with neurological disorders (e.g., multiple sclerosis, Parkinson's disease).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | monitored through 36 months post-treatment
  rate of adverse events reported for each patient

SECONDARY OUTCOMES:
Number of participants with graft thrombosis or grant failures | monitored through 36 months post-treatment
  lack of graft thrombosis or graft failure

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P Terlecki, MD, Principal Investigator — Associate Professor
Locations (1):
- Wake Forest Institute for Regenerative Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No